CLINICAL TRIAL: NCT01274169
Title: Measurment of GFR by Nasal Sensors
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Ministry of health israel, Ministry of health israel
Other Study IDs: NANOCTIL
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2008-02

CONDITIONS: Measure GFR by Nasal Sensor

SUMMARY:
to measure kidney function by measuring blood creatinine and to compare it to the measurment of GFR by Nanotechnology

ELIGIBILITY:
Inclusion Criteria:

adults between 18-70 yrs

Exclusion Criteria:

subject under 18

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: volunteers subjects with different stages of CKD
Sampling Method: Non-Probability Sample
Dates: Start 2008-03; Study Completion 2010-03